CLINICAL TRIAL: NCT05220982
Title: Improving Efficacy of Voice Therapy Concepts Via Telepractice and Mobile App Technology
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West Chester University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R15DC019954 (NIH)
Record Dates: First submitted 2022-01-06; First posted 2022-02-02 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Voice Disorders
MeSH Terms: conditions — Voice Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Conversation Training Therapy (Experimental)
  Interventions: Behavioral: Conversation Training Therapy
- Global Voice Prevention and Therapy Model (Experimental)
  Interventions: Behavioral: Global Voice Prevention and Therapy Model
- Modified Conversation Training Therapy (Experimental)
  Interventions: Behavioral: Modified Conversation Training Therapy
- Modified Global Voice Prevention and Therapy Model (Experimental)
  Interventions: Behavioral: Modified Global Voice Prevention and Therapy Model

INTERVENTIONS:
Behavioral: Conversation Training Therapy — Training clear speech in conversation with new vs old voice. Training will occur over four weekly synchronous telepractice sessions. Each session lasts 45-60 minutes. The ecological momentary intervention (EMI) platform (app, server, web portal) will reflect the goals of the intervention. Participants will use the EMI platform to practice voice targets three times a day.
  Arms: Conversation Training Therapy
Behavioral: Global Voice Prevention and Therapy Model — Training of four new voices (i.e., resonant voice in connected speech, falsetto for quiet talking, oral twang for talking over noise, and belt for healthy yelling) defined and trained by the anatomy and physiology of the system (i.e., Estill Voice Training's Figures). Training occurs in a bottom-up speech hierarchy with new vs other or old voice at each step. Additional methods are used in asynchronous telepractice to support the new voices during week 1 (e.g., vocal hygiene and education). Training will occur over three weekly synchronous telepractice sessions. Each session lasts 45-60 minutes. The ecological momentary intervention (EMI) platform (app, server, web portal) will reflect the goals of the intervention. Participants will use the EMI platform to practice voice targets three times a day.
  Arms: Global Voice Prevention and Therapy Model
Behavioral: Modified Conversation Training Therapy — Training clear speech in conversation with no use of new vs old voice. Training will occur over four weekly synchronous telepractice sessions. Each session lasts 45-60 minutes. The ecological momentary intervention (EMI) platform (app, server, web portal) will reflect the goals of the intervention. Participants will use the EMI platform to practice voice targets three times a day.
  Arms: Modified Conversation Training Therapy
Behavioral: Modified Global Voice Prevention and Therapy Model — Training of a new resonant voice in connected speech defined and trained by the anatomy and physiology of the system (i.e., Estill Voice Training's Figures). Training occurs in a bottom-up speech hierarchy with no use of new vs old voice. Additional methods are used in asynchronous telepractice to support the new voices during week 1 (e.g., vocal hygiene and education). Training will occur over three weekly synchronous telepractice sessions. Each session lasts 45-60 minutes. The ecological momentary intervention (EMI) platform (app, server, web portal) will reflect the goals of the intervention. Participants will use the EMI platform to practice voice targets three times a day.
  Arms: Modified Global Voice Prevention and Therapy Model

SUMMARY:
Due to the COVID-19 pandemic, telepractice has grown rapidly. To date, synchronous telepractice (i.e., in real-time videoconferencing) has been the focus of most research with asynchronous telepractice (i.e. information stored and accessed later) being used minimally only to record synchronous encounters. Descriptions of voice therapy concepts are minimally available in the literature with no standard reporting framework and no clinical efficacy or effectiveness data. Thus, the proposed study will address these barriers. First, an asynchronous method will be developed that will impact both in-person and telepractice services by offering repeated learning opportunities in the client's environment. The method includes ecological momentary intervention (EMI) through a daily voice therapy practice app, server, and web portal that is flexible in its programming to meet the needs of the client, offers performance feedback, and charts results over time. Second, voice therapy concepts will be tested improving our knowledge about such concepts that facilitate successful client-centered outcomes for both prevention and treatment of voice problems. The participants in the study will be teachers who have a high prevalence of voice problems, impact the healthcare system when treatment is needed, and negatively affect students' learning abilities in the classroom when communicating with a voice problem. Third, the Rehabilitation Treatment Specification System (RTSS) framework will be used to describe the voice therapy concepts. The concepts include: training multiple voices to meet all the clients' vocal needs, defining voice qualities by the anatomy and physiology of the voice production system, generalizing voice targets into hierarchical speech tasks, and using "new" vs "other/old" voice to help the client become their own clinician. Vocally healthy student teachers and professional teachers with voice complaints will be randomized into one of four voice therapy conditions delivered via telepractice. Both groups of teachers are needed to assess the concepts for prevention and treatment. Condition 2, which fully represents the proposed voice therapy concepts, will be superior to the other three conditions, which do not fully represent the concepts, by demonstrating a greater decrease in client-reported primary outcome measures of the Voice Handicap Index-10 and factor 1 and 2 of the Vocal Fatigue Index. Secondary outcomes of acoustic measures, Borg Category Ratio-10 scales for vocal and mental effort, and voice therapy satisfaction surveys will also be investigated. The results will be useful at a practical level by advancing asynchronous telepractice and by improving efficacy of voice therapy concepts. In addition, the results will lay the groundwork for future studies involving development of EMI platforms in other areas of speech-language pathology and testing additional voice therapy concepts that facilitate successful client-centered outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Vocally healthy student in a bachelor of education program with student teaching planned for spring
* Professional teacher who is currently working as a teacher with voice complaints, but has not sought help for the complaints
* Owner of either an android or iOS smartphone or tablet.

Exclusion Criteria:

* Not a student teacher
* Not a professional teacher.
* Does not own a smartphone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-08-31 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Voice Handicap Index 10 | One time at pre & one time at post condition in fall (4 weeks between pre and post) and once weekly for 15 weeks in spring. Captured on day 4 in the PM for a 5 day period via the VoiceEvalU8 app.
  The VHI-10 is a client reported outcome measure related to voice impact on quality of life across 10 questions. Each question is rated on a scale from 0-4 with 0 as never, 1 as almost never, 2 as sometimes, 3 as almost always, and 4 as always.
Change in Vocal Fatigue Index (VFI) factor 1 and 2 | One time at pre & one time at post condition in fall (4 weeks between pre and post) and once weekly for 15 weeks in spring. Captured on day 5 in the PM for a 5 day period via the VoiceEvalU8 app.
  The VFI is a client reported outcome measure related to tiredness and avoidance of voice in factor 1 and physical voice discomfort in factor 2. Factor 1 has 11 questions and factor 2 has 5 questions. Each question is rated on a scale from 0-4 with 0 as never, 1 as almost never, 2 as sometimes, 3 as almost always, and 4 as always.

SECONDARY OUTCOMES:
Change in Fundamental Frequency | One time at pre & one time at post condition in fall (4 weeks between pre and post) and weekly for 15 weeks in spring. Captured twice a day in AM and PM sessions during a 5 day period via the VoiceEvalU8 app.
  Fundamental frequency will be measured during 3 trials of 5-sec sustained /a/s, the phrase, "we were away a year ago," and a 15-sec connected speech sample.
Change in Jitter% | One time at pre & one time at post condition in fall (4 weeks between pre and post) and weekly for 15 weeks in spring. Captured twice a day in AM and PM sessions during a 5 day period via the VoiceEvalU8 app.
  Jitter% will be measured during 3 trials of 5-sec sustained /a/s, the phrase, "we were away a year ago," and a 15-sec connected speech sample.
Change in noise-to-harmonic ratio | One time at pre & one time at post condition in fall (4 weeks between pre and post) and weekly for 15 weeks in spring. Captured twice a day in AM and PM sessions during a 5 day period via the VoiceEvalU8 app.
  Noise-to-harmonic ratio will be measured during 3 trials of 5-sec sustained /a/s, the phrase, "we were away a year ago," and a 15-sec connected speech sample.
Change in cepstral peak prominence | One time at pre & one time at post condition in fall (4 weeks between pre and post) and weekly for 15 weeks in spring. Captured twice a day in AM and PM sessions during a 5 day period via the VoiceEvalU8 app.
  Cepstral peak prominence will be measured during 3 trials of 5-sec sustained /a/s, the phrase, "we were away a year ago," and a 15-sec connected speech sample.
Change in smoothed cepstral peak prominence | One time at pre & one time at post condition in fall (4 weeks between pre and post) and weekly for 15 weeks in spring. Captured twice a day in AM and PM sessions during a 5 day period via the VoiceEvalU8 app.
  Smoothed cepstral peak prominence will be measured during 3 trials of 5-sec sustained /a/s, the phrase, "we were away a year ago," and a 15-sec connected speech sample.
Change in acoustic voice quality index | One time at pre & one time at post condition in fall (4 weeks between pre and post) and weekly for 15 weeks in spring. Captured twice a day in AM and PM sessions during a 5 day period via the VoiceEvalU8 app.
  Acoustic voice quality index will be measured during 1 trial of the 5-sec sustained /a/ and the phrase, "we were away a year ago,"
Change in Borg Category Ratio (CR)10 scale for vocal effort | One time at pre & one time at post condition in fall (4 weeks between pre and post) and weekly for 15 weeks in spring. Captured once a day in PM sessions during a 5 day period via the VoiceEvalU8 app.
  The Borg CR10 scale rates vocal effort on a scale from 0-10 with 0 as no effort and 10 as maximum effort.
Change in Borg Category Ratio (CR)10 scale for mental effort | One time at pre & one time at post condition in fall (4 weeks between pre and post) and weekly for 15 weeks in spring. Captured once a day in PM sessions during a 5 day period via the VoiceEvalU8 app.
  The Borg CR10 scale rates mental effort on a scale from 0-10 with 0 as no effort and 10 as maximum effort.
Student researcher (SR) voice therapy satisfaction surveys | Collected immediately after intervention in the fall via Qualtrics online software.
  The voice therapy satisfaction survey will rate the student researchers' (SR) perceptions after completing the voice therapy conditions. The questions are rated on a scale from 1-5 with 1 as strongly disagree and 5 as strongly agree.
  There are also some open ended responses. The SR survey has 17 questions.
Participant voice therapy satisfaction surveys | Collected immediately after intervention in the fall via Qualtrics online software.
  The voice therapy satisfaction surveys will rate the participants' perceptions after completing the voice therapy conditions. The questions are rated on a scale from 1-5 with1 as strongly disagree and 5 as strongly agree.
  There are also some open ended responses. The participant survey has 12 questions.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth U Grillo, Ph.D., Principal Investigator — West Chester University
Locations (1):
- Elizabeth Grillo, West Chester, Pennsylvania, United States